CLINICAL TRIAL: NCT00001314
Title: Investigation of Myocardial Contractile Reserve by Dobutamine Stress Transesophageal Echocardiography in Aortic and Mitral Regurgitation
Brief Title: Investigation of Heart Function in Patients With Heart Valve Defects
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 920195; 92-H-0195
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-04

CONDITIONS: Aortic Valve Insufficiency; Mitral Valve Insufficiency
Keywords: Aortic Regurgitation; Dobutamine Stress; Left Ventricular Function; Mitral Regurgitation; Myocardial Contractile Reserve; Transesophageal Echocardiography
MeSH Terms: conditions — Aortic Valve Insufficiency; Mitral Valve Insufficiency

SUMMARY:
In this study researchers plan to perform a diagnostic test called transesophageal echocardiography in order to see and record the movement and function of the heart.

Transesophageal echocardiography is similar to an upper gastrointestinal endoscopy. Different views of the heart are taken by a small, flexible instrument positioned in the esophagus (the tube that connects the mouth to the stomach). This allows doctors to create a clear picture of the heart through the wall of the esophagus rather than from outside the body through the muscles, fat, and bones of the chest wall.

During transesophageal echocardiography pictures of the heart will be taken while patients rest and as patients receive a medication called dobutamine. Dobutamine is a medication that makes the heart beat stronger and faster, similar to what exercise does to the heart.

Researchers are particularly interested in studying patients with defects in the valves of the heart, especially aortic regurgitation and mitral regurgitation. Patients with these defects in the heart valves tend to develop abnormalities in the size and function of the left ventricle. The left ventricle is one of the four chambers of the heart responsible for ejecting blood out of the heart into the circulation. Researchers believe that by identifying changes in the function of heart muscle, they may be able to predict the occurrence of muscle damage due to the diseased valves.

The purpose of this study is to determine whether the function of heart muscle measured during dobutamine stress transesophageal echocardiography can predict the later development of problems in the function and size of the left ventricle.

DETAILED DESCRIPTION:
In this investigation, we propose to perform dobutamine stress transesophageal echocardiography in patients with aortic regurgitation and in patients with mitral regurgitation in order to assess myocardial contractile reserve. The purpose of the study is to determine whether the contractile reserve of the myocardium measured during dobutamine stress echocardiography is a predictor of the development of subsequent left ventricular dysfunction and left ventricular dilatation, as well as recovery of left ventricular function after surgery, in these patients.

ELIGIBILITY:
18 - 65 years of age.

Patients with severe aortic regurgitation and patients with severe mitral regurgitation.

Patients will discontinue medications 48 hours prior to the study.

Women must not be pregnant.

Patients must not have an associated valvular heart disease (i.e., patients with aortic regurgitation will be excluded if there is coexistent mitral valve disease; patients with mitral regurgitation will be excluded if there is coexistent aortic valve disease).

Patients must not have any form of cardiomyopathy.

Patients must not have coronary artery disease.

Patients must not have ventricular ectopy during baseline conditions (i.e., couplets, frequent PVc's [greater than 6/min], early coupling ["R-on-T" phenomenon], ventricular bigeminy) that might potentially predispose the patient for the development of dangerous dysrhythmia during dobutamine infusion.

Patients must not have a history of cardiac arrest or ventricular tachycardia.

Patients must not have a history of congestive heart failure.

Patients must not have hypotension (i.e., systolic blood pressure less than 100 mmHg).

Patients must not have a systolic blood pressure greater than 200 mmHg.

Patients must not have a left atrial size of greater than 100 mm.

Patients must not have atrial fibrillation.

Patients must not have sinus tachycardia greater than or equal to 100 beats/min.

Patients must not have esophageal disease.

Patients must not have any other medical condition that , at the discretion of the physician in charge, may increase the risk of the procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 1992-05; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Ross J Jr. Afterload mismatch in aortic and mitral valve disease: implications for surgical therapy. J Am Coll Cardiol. 1985 Apr;5(4):811-26. doi: 10.1016/s0735-1097(85)80418-6. PMID 3882814
- [Background] Bonow RO, Rosing DR, McIntosh CL, Jones M, Maron BJ, Lan KK, Lakatos E, Bacharach SL, Green MV, Epstein SE. The natural history of asymptomatic patients with aortic regurgitation and normal left ventricular function. Circulation. 1983 Sep;68(3):509-17. doi: 10.1161/01.cir.68.3.509. No abstract available. PMID 6872164
- [Background] Bonow RO, Lakatos E, Maron BJ, Epstein SE. Serial long-term assessment of the natural history of asymptomatic patients with chronic aortic regurgitation and normal left ventricular systolic function. Circulation. 1991 Oct;84(4):1625-35. doi: 10.1161/01.cir.84.4.1625. PMID 1914102